CLINICAL TRIAL: NCT02248480
Title: Effect of Duloxetine 60 mg Versus Placebo in Patients With Chronic Osteoarthritis and Knee Pain in Japan
Brief Title: A Study of Duloxetine (LY248686) in Participants With Chronic Osteoarthritis and Knee Pain in Japan
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Collaborators: Shionogi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 14375; F1J-JE-HMGX (Other: Eli Lilly and Company)
Record Dates: First submitted 2014-09-22; First posted 2014-09-25 (Estimated); Results first posted 2017-01-16 (Estimated); Last update posted 2019-09-26 (Actual); Status verified 2019-09

CONDITIONS: Osteoarthritis of the Knee
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Duloxetine Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Duloxetine (Experimental): Duloxetine 20 milligram (mg) for first week, 40 mg for second week and 60 mg for next 12 weeks administered orally once daily. Tapering week doses of 40 mg for three days and 20 mg for four days.
  Interventions: Drug: Duloxetine
- Placebo (Placebo Comparator): Placebo administered orally once a day for 15 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Duloxetine — Administered orally
  Other Names: LY248686
  Arms: Duloxetine
Drug: Placebo — Administered orally
  Arms: Placebo

SUMMARY:
The main purpose of this study is to evaluate the efficacy of the study drug known as duloxetine in participants with chronic osteoarthritis (OA) and knee pain in Japan.

ELIGIBILITY:
Inclusion Criteria:

* Participants with present OA.
* Have pain for ≥ 14 days of each month for 3 months prior to study entry.
* Participants must have a score of ≥4 on the BPI average pain score before randomization.
* Females of child-bearing potential must test negative (-) on a pregnancy test.

Exclusion Criteria:

* Participants who cannot appropriately complete the daily diaries.
* Have a score change of ≧3 on BPI 24-hour average pain score between screening and baseline.
* Participants who have serious cardiovascular, hepatic, renal, endocrine, respiratory, or hematologic illness, peripheral vascular disease, or other medical condition or neuropsychiatric conditions or clinically significant laboratory abnormalities or electrocardiographic abnormalities.
* Participants who have alanine aminotransferase (ALT) or aspartate aminotransferase (AST) higher than 100 international units per liter (IU/L) or total bilirubin higher than 1.6 milligrams/deciliter (mg/dL).
* Participants who have serum creatinine level higher than 2.0 mg/dL, or had renal transplantation or are receiving renal dialysis.
* Participants who have a diagnosis of inflammatory arthritis (that is, rheumatoid arthritis) or an autoimmune disorder (excluding inactive Hashimoto's thyroiditis and Type 1 diabetes).
* Participants who have any previous diagnosis of psychosis, bipolar disorder, or schizoaffective disorder.
* Participants who have major depressive disorder as determined using depression module of the Mini-International Neuropsychiatric Interview (M.I.N.I.).
* Participants who have uncorrected thyroid disease, uncontrolled narrow-angle glaucoma, history of uncontrolled seizures, or uncontrolled or poorly controlled hypertension.
* Participants who have received intrarticular hyaluronate or steroids, joint lavage, or other invasive therapies to the knee in the past 1 month.
* Participants who have had knee arthroscopy of the index knee within the past year or joint replacement of the index knee or osteotomy at anytime.
* Participants who have end-stage osteoarthritis or surgery planned during the trial for the index joint.
* Participants have a prior synovial fluid analysis showing a white blood cell (WBC) ≥2000 cubic millimeters (mm3) that is indicative of a diagnosis other than OA.
* Participants taking any excluded medications that cannot be discontinued.
* Participants anticipated by the investigator to require use of nonsteroidal anti-inflammatory drugs that include acetaminophen, opioid analgesics, or other excluded medication for the duration of the study.
* Participants treated with a monoamine oxidase inhibitor (MAoI) within 14 days prior to baseline, or those with the potential need to use MAO inhibitor during the study or within 5 days of discontinuation of investigational drug.
* Participants who answer 'yes' to any of the questions about active suicidal ideation/intent/behaviors occurring within the past month (Columbia-Suicide Severity Rating Scale, suicide ideation section-questions 4 and 5; suicidal behaviors section).
* Participants who have a history of having more than one medical allergy.
* Are non-ambulatory or require the use of crutches or a walker.
* Have frequent falls that could result in hospitalization or could compromise response to treatment.
* Have a primary painful condition that may interfere with assessment of the index joint, i.e., knee.
* Have a history of drug abuse or dependence within the past year, including alcohol and excluding nicotine and caffeine.
* Have a positive urine drug screen for any substances of abuse or excluded medication.
* Have received administration of another investigational drug within the 30 days prior to screening.
* Have had previous exposure to duloxetine or completed/withdrawn from any study investigating duloxetine.
* Pregnant participants, female participants who wish to be pregnant during the clinical study period, or participants who are breast-feeding; or male participants who wish pregnancy of the partner.

Ages: 40 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 354 (Actual)
Dates: Start 2014-10; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hyōgo, Japan

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

REFERENCES:
- [Derived] Leaney AA, Lyttle JR, Segan J, Urquhart DM, Cicuttini FM, Chou L, Wluka AE. Antidepressants for hip and knee osteoarthritis. Cochrane Database Syst Rev. 2022 Oct 21;10(10):CD012157. doi: 10.1002/14651858.CD012157.pub2. PMID 36269595
- [Derived] Itoh N, Tsuji T, Ishida M, Ochiai T, Konno S, Uchio Y. Efficacy of duloxetine for multisite pain in patients with knee pain due to osteoarthritis: An exploratory post hoc analysis of a Japanese phase 3 randomized study. J Orthop Sci. 2021 Jan;26(1):141-148. doi: 10.1016/j.jos.2020.02.013. Epub 2020 Mar 31. PMID 32245696
- [Derived] Enomoto H, Fujikoshi S, Ogawa K, Tsuji T, Tanaka S. Relationship Between Pain Reduction and Improvement in Health-Related Quality of Life in Patients with Knee Pain Due to Osteoarthritis Receiving Duloxetine: Exploratory Post Hoc Analysis of a Japanese Phase 3 Randomized Study. J Pain Res. 2020 Jan 20;13:181-191. doi: 10.2147/JPR.S211072. eCollection 2020. PMID 32021407
- [Derived] Yue L, Wang J, Enomoto H, Fujikoshi S, Alev L, Cheng YY, Skljarevski V. The Clinical Relevance of Pain Severity Changes: Is There Any Difference Between Asian and Caucasian Patients With Osteoarthritis Pain? Pain Pract. 2020 Feb;20(2):129-137. doi: 10.1111/papr.12835. Epub 2019 Nov 20. PMID 31505082
- [Derived] Itoh N, Tsuji T, Ishida M, Ochiai T, Konno S, Uchio Y. Response to duloxetine in patients with knee pain due to osteoarthritis: an exploratory post hoc analysis of a Japanese Phase III randomized study. J Pain Res. 2018 Oct 26;11:2603-2616. doi: 10.2147/JPR.S176036. eCollection 2018. PMID 30464579
- [Derived] Enomoto H, Fujikoshi S, Tsuji T, Sasaki N, Tokuoka H, Uchio Y. Efficacy of duloxetine by prior NSAID use in the treatment of chronic osteoarthritis knee pain: A post hoc subgroup analysis of a randomized, placebo-controlled, phase 3 study in Japan. J Orthop Sci. 2018 Nov;23(6):1019-1026. doi: 10.1016/j.jos.2018.07.008. Epub 2018 Aug 17. PMID 30126675
- [Derived] Uchio Y, Enomoto H, Alev L, Kato Y, Ishihara H, Tsuji T, Ochiai T, Konno S. A randomized, double-blind, placebo-controlled Phase III trial of duloxetine in Japanese patients with knee pain due to osteoarthritis. J Pain Res. 2018 Apr 18;11:809-821. doi: 10.2147/JPR.S164128. eCollection 2018. PMID 29713194

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: All started participants (pt) were randomized and received at least one dose of study drug. Efficacy population had at least 1 post-dose efficacy assessment.
Period: Overall Study
Arm/Group | Duloxetine | Placebo
Started | 178 | 176
Efficacy Population | 177 | 176
Completed | 161 | 162
Not Completed | 17 | 14
Not completed — Lack of Efficacy | 4 | 6
Not completed — Adverse Event | 11 | 2
Not completed — Withdrawal by Subject | 2 | 4
Not completed — Entry Criteria Not Met | 0 | 1
Not completed — Other:Physician Decision | 0 | 1

BASELINE CHARACTERISTICS:
Population: Al randomized participants who received at least 1 dose of study drug and had 1 post-dose efficacy assessment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Duloxetine | Placebo | Total
Number analyzed (Participants) | 177 | 176 | 353
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.5 (8.0) | 66.4 (8.4) | 65.9 (8.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 142 | 132 | 274
  Male | 35 | 44 | 79
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 177 | 176 | 353
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Japan | 177 | 176 | 353

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline on the Brief Pain Inventory (BPI) 24-Hour Average Pain Score
Description: Brief Pain Inventory Severity: Average Pain Score: A self-reported scale that measures the severity of pain based on the average pain experienced during the past 24-hours. The severity scores ranged from 0 (no pain) to 10 (pain as severe as you can imagine). Least squares (LS) mean was calculated using a mixed-effects model repeated measures (MMRM) approach including administration groups, observation points, and interaction between the administration groups and observation points as fixed effects, and BPI average pain severity at baseline as covariates.
Time Frame: Baseline, Week 14
Population: All randomized participants who received at least 1 dose of study drug and had at least 1 post-dose efficacy assessment.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 177 | 176
units on a scale | -2.57 (0.12) | -1.80 (0.12)
Statistical Analysis 1: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p < .0001, Mixed Models Analysis

2. Secondary Outcome: Change From Baseline in Patient Global Impression of Improvement (PGI-Improvement)
Description: Patient's Global Impressions of Improvement Scale: PGI-I measures a participant's perception of improvement at the time of assessment compared with the start of treatment. Score ranges from 1 (very much better) to 7 (very much worse). Least squares (LS) mean was calculated using a mixed-effects model repeated measures (MMRM) approach including administration groups, observation points, and interaction between the administration groups and observation points as fixed effects, and PGI-severity at baseline as covariates.
Time Frame: Baseline, 14 Weeks
Population: All randomized participants who received at least 1 dose of study drug and had at least 1 post-dose efficacy assessment.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 177 | 176
units on a scale | 2.23 (0.09) | 2.84 (0.09)

3. Secondary Outcome: Change From Baseline on the Clinical Global Impression of Severity (CGI-S)
Description: CSI-S measures severity of illness at the time of assessment compared with start of treatment with scores ranging from 1 (normal, not at all ill) to 7 (among the most extremely ill participants). Least squares (LS) mean was calculated using a mixed-effects model repeated measures (MMRM) approach including administration groups, observation points, and interaction between the administration groups and observation points as fixed effects, and baseline data as covariates.
Time Frame: Baseline, Week 14
Population: All randomized participants who received at least 1 dose of study drug and had at least 1 post-dose efficacy assessment.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 177 | 176
units on a scale | -1.71 (0.07) | -1.22 (0.07)

4. Secondary Outcome: Change From Baseline on the 36-Item Short-Form Health Survey (SF-36)
Description: 36-item Short-Form Health Survey: SF-36 Health Status Survey is a generic, health-related scale assessing participant's quality of life on 8 domains: physical functioning, social functioning, bodily pain, vitality, mental health, role-physical, role-emotional and general health. Domain scores: general health (range: 5-25); physical functioning (range: 10-30); role-physical (range: 4-8); role-emotional (range: 3-15); social functioning (range: 2-10); bodily pain (range: 2-12); vitality (range: 4-20); mental health (range: 5-25). Each raw scale score was converted to a scale score ranging from 0-100 points, , with higher values representing a better outcome [(Raw score) - min{raw score}] / (max {raw score} - min{raw score}) x 100]. Least squares (LS) mean was calculated using Analysis of covariance (ANCOVA) approach including administration groups as fixed effects, and baseline data as covariate.
Time Frame: Baseline, Week 14
Population: All participants who received at least 1 dose of study drug and had at least 1 post-dose efficacy assessment. The last observation carried forward (LOCF) was used.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 177 | 176
units on a scale
  Physical Functioning | 12.62 (1.27) | 6.23 (1.27)
  Role (Physical) | 11.44 (1.29) | 3.66 (1.30)
  Bodily Pain | 16.32 (1.22) | 9.63 (1.22)
  General Health | 5.58 (0.93) | 1.82 (0.94)
  Vitality | 3.99 (1.04) | 3.16 (1.04)
  Social Functioning | 5.66 (1.14) | 2.54 (1.15)
  Role (Emotional) | 6.32 (1.27) | 0.70 (1.28)
  Mental Health | 3.02 (0.99) | 1.48 (0.99)

5. Secondary Outcome: Change From Baseline on the Beck Depression Inventory (BDI-II) Total Score
Description: Beck Depression Inventory-II: BDI-II is a 21-item, participant-completed questionnaire to assess characteristics of depression. Each of the 21 items corresponding to symptoms of depression were scored on a 4-point scale ranging from 0 to 3 and was summed to give a single score. A total score of 0-13 was considered minimal range, 14-19 was mild, 20-28 was moderate, and 29-63 was severe. Least squares (LS) mean was calculated using a ANCOVA approach' including administration groups as fixed effects, and baseline data as covariate.
Time Frame: Baseline, Week 14
Population: All randomized participants who received at least 1 dose of study drug and had at least 1 post-dose efficacy assessment. The last observation carried forward (LOCF) was used.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 177 | 176
units on a scale | -0.78 (0.23) | -0.51 (0.24)

6. Secondary Outcome: Percentage of Participants With Fall Events From Fall Questionnaire
Description: Participants evaluated their experience with and details of falls which were recorded.
Time Frame: Baseline through Week 14
Population: All randomized participants who received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 178 | 176
percentage of participants | 10.1 | 9.7

7. Secondary Outcome: Change From Baseline on the Western Ontario and McMaster Osteoarthritis Index (WOMAC) Questionnaire Total Score
Description: The 24-question WOMAC Osteoarthritis Index assesses osteoarthritis symptoms using pain (5 questions), stiffness (2 questions) and physical function (17 questions) subscales. The WOMAC Osteoarthritis Index version 3.1 was administered according to the study schedule. The WOMAC total score was calculated for each participant at each time point for analysis as the mean total score, range 0 (none) -96 (extreme). Least squares (LS) mean was calculated using a mixed-effects model repeated measures (MMRM) approach including administration groups, observation points, and interaction between the administration groups and observation points as fixed effects, and baseline data as covariates.
Time Frame: Baseline, Week 14
Population: All randomized participants who received at least 1 dose of study drug and had at least 1 post-dose efficacy assessment.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 177 | 176
units on a scale | -17.41 (0.91) | -10.45 (0.91)

8. Secondary Outcome: Change From Baseline on the Patient Global Assessment Illness (PGAI) Score
Time Frame: Baseline, Week 14
Population: Zero participants analyzed. PGAI outcome measure was registered incorrectly thus no analysis produced.
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Change From Baseline on the 5 Dimension (EQ-5D) Version of the European Quality of Life Instrument
Description: The EQ-5D is a generic, multidimensional, health-related, quality-of-life instrument and was completed on five dimensions (mobility, self care, usual activities, pain/discomfort and anxiety/depression) to measure health-related quality of life on a scale from 0-1, with the higher score indicating a better health state perceived by the participant. The profile allows participants to rate their health state in 5 health domains: mobility, self-care, usual activities, pain/discomfort, and mood using a three level scale (no problem, some problems, and major problems). These combinations of attributes were converted into a weighted health-state Index Score according to the Japan population-based algorithm. Least squares (LS) mean was calculated using an ANCOVA approach including administration groups as fixed effects, and baseline data as covariate.
Time Frame: Baseline, Week 14
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 177 | 176
units on a scale | 0.12 (0.01) | 0.07 (0.01)

10. Secondary Outcome: Change in Baseline in Brief Pain Inventory Severity and Interference Scores (BPI-S, BPI-I) Change From Baseline in BPI Pain Severity Items and Interference Items Score
Description: BPI-S and BPI-I are self-reported scales measuring severity of pain and interference on function. Severity scores: 0 (no pain) to 10 (severe pain) on each question assessing worst pain, least pain, and average pain in past 24 hours, and pain right now. Interference scores: 0 (does not interfere) to 10 (completely interferes) on each question assessing interference of pain in past 24 hours for general activity, mood, walking ability, normal work, relations with other people, sleep, and enjoyment of life. Average interference = average of non-missing scores of individual interference items. Least squares (LS) mean was calculated using a mixed-effects model repeated measures (MMRM) approach including administration groups, observation points, and interaction between the administration groups and observation points as fixed effects, and baseline data as covariates.
Time Frame: Baseline, Week 14
Population: All randomized participants who received at least 1 dose of study drug and had at least 1 post-dose efficacy assessment.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 177 | 176
units on a scale
  Worse Pain | -2.92 (0.15) | -2.13 (0.15)
  Least Pain | -1.61 (0.11) | -1.05 (0.11)
  Pain Right Now | -2.29 (0.13) | -1.52 (0.13)
  General Activity | -2.42 (0.14) | -1.52 (0.14)
  Walking Ability | -2.58 (0.14) | -1.74 (0.14)
  Mood | -1.95 (0.12) | -1.43 (0.12)
  Normal Work | -2.48 (0.13) | -1.67 (0.13)
  Relationship to People | -1.23 (0.11) | -0.81 (0.11)
  Sleep | -1.65 (0.11) | -1.19 (0.11)
  Enjoyment of Life | -1.78 (0.12) | -1.16 (0.12)
  Average of 7 Items | -2.01 (0.11) | -1.34 (0.11)

11. Secondary Outcome: Percentage of Participants With a 30% and 50% Reduction in Average Pain Score on Weekly Mean of the 24-Hour Average Pain Score on the 11-Point Numeric Rating Scale
Description: 24-hour average pain severity scores were recorded daily on an 11-point Likert scale, an ordinal scale, with scores ranging from 0 (no pain) to 10 (worst possible pain). The 11-point Likert scale was also used for assessment of average pain within 24-hours.
Time Frame: Baseline,Week 14
Population: as for outcome 5
Measure: Number; unit: percentage of participants
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 177 | 176
percentage of participants
  >=30% | 72.3 | 52.8
  >=50% | 55.4 | 38.6

12. Secondary Outcome: Change From Baseline on Weekly Mean of the 24-Hour Average Pain and Worst Pain Score
Description: 24-hour average pain severity scores were recorded daily on an 11-point Likert scale, an ordinal scale, with scores ranging from 0 (no pain) to 10 (worst possible pain). The 11-point Likert scale was also used for assessment of average pain and worst pain within 24-hours. Least squares (LS) mean was calculated using a mixed-effects model repeated measures (MMRM) approach including administration groups, observation points, and interaction between the administration groups and observation points as fixed effects, and baseline data as covariates.
Time Frame: Baseline, Week 14
Population: All randomized participants who received at least 1 dose of study drug and had at least 1 post-dose efficacy assessment.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 177 | 176
units on a scale
  Average Pain | -2.45 (0.12) | -1.79 (0.12)
  Worst Pain | -2.73 (0.14) | -1.97 (0.14)

13. Secondary Outcome: Percentage of Participants With Reduction of ≥30% and ≥50% in BPI Average Pain Score
Description: Brief Pain Inventory Severity: Average Pain Score: A self-reported scale that measures the severity of pain based on the average pain experienced during the past 24-hours. The severity scores ranged from 0 (no pain) to 10 (pain as severe as you can imagine).
Time Frame: Baseline, Week 14
Population: as for outcome 5
Measure: Number; unit: percentage of participants
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 177 | 176
percentage of participants
  >=30% | 72.3 | 52.8
  >=50% | 55.4 | 38.6

14. Secondary Outcome: Percentage of Participants With a Responder Rate Based on OMERACT-OARSI Criteria
Description: A responder is required to meet at least one condition: reduction of ≥50% and ≥2 score in Weekly Mean of the 24-Hour Average Pain Score, reduction of ≥50% or ≥13.6 score in WOMAC (difficulty in dairy activity) and meet ≥2 out of following 3 conditions: reduction of ≥20% and ≥1 score in Weekly Mean of the 24-Hour Average Pain, reduction of ≥20% and ≥6.8 score in WOMAC (difficulty in dairy activity), PGAI score ≥2.
Time Frame: Baseline, Week 14
Population: as for outcome 5
Measure: Number; unit: percentage of participants
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 177 | 176
percentage of participants | 83.6 | 61.9

15. Secondary Outcome: Change From Baseline on the WOMAC Questionnaire Pain Subscale
Description: The WOMAC index (pain, stiffness, physical function subscales) was completed by the participant.The pain subscale had 5 questions on pain associated with every day tasks. Each question was answered using a 5-point Likert scale (0 to 4). The pain subscale has a range of scores of 0 (none) to 20 (extreme). Least squares (LS) mean was calculated using a mixed-effects model repeated measures (MMRM) approach including administration groups, observation points, and interaction between the administration groups and observation points as fixed effects, baseline data as covariates.
Time Frame: Baseline, 14 Weeks
Population: All randomized participants who received at least 1 dose of study drug and had at least 1 post-dose efficacy assessment.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 177 | 176
units on a scale | -3.99 (0.21) | -2.43 (0.21)

16. Secondary Outcome: Change From Baseline on the WOMAC Questionnaire Stiffness Subscale
Description: The WOMAC index (pain, stiffness, physical function subscales) will be completed by the participant.The stiffness subscale had 2 questions on stiffness associated with time of day (morning versus later in the day). Each question was answered using a 5-point Likert scale (0 to 4). The stiffness subscale has a range of scores of 0 (none) to 8 (extreme). Least squares (LS) mean was calculated using a mixed-effects model repeated measures (MMRM) approach including administration groups, observation points, and interaction between the administration groups and observation points as fixed effects, baseline data as covariates.
Time Frame: Baseline, 14 Weeks
Population: All randomized participants who received at least 1 dose of study drug and had at least 1 post-dose efficacy assessment.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 177 | 176
units on a scale | -1.66 (0.09) | -0.98 (0.09)

17. Secondary Outcome: Change From Baseline on the WOMAC Questionnaire Physical Function Subscale
Description: The WOMAC osteoarthritis scale consists of 24 items in 3 subscales: pain, stiffness, and physical function. The physical function subscale rates participant pain during stair use, rising from sitting, standing, bending, walking, getting in/out of a car, shopping, putting on/taking off socks, rising from bed, lying in bed, getting in/out of the bath, sitting, getting on/off the toilet, heavy household duties, and light household duties. Each question was answered using a 5-point Likert scale (0 to 4). Physical Function Subscale has a range of scores of 0 (none) to 68 (extreme). Least squares (LS) mean was calculated using a mixed-effects model repeated measures (MMRM) approach including administration groups, observation points, and interaction between the administration groups and observation points as fixed effects, baseline data as covariates.
Time Frame: Baseline, 14 Weeks
Population: All randomized participants who received at least 1 dose of study drug and had at least 1 post-dose efficacy assessment.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 177 | 176
units on a scale | -11.77 (0.67) | -7.07 (0.66)

ADVERSE EVENTS:
Description: All randomized participants who received at least 1 dose of study drug.
Arm/Group | Duloxetine | Placebo
Serious Adverse Events (participants affected / at risk) | 1/178 | 1/176
Other Adverse Events (participants affected / at risk) | 120/178 | 98/176
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Duloxetine (N=178) | Placebo (N=176)
Cerebellar tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Malignant ascites (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Duloxetine (N=178) | Placebo (N=176)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0)
Ear congestion (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 2 (2) | 2 (2)
Vertigo positional (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Basedow's disease (Endocrine disorders) | 1 (1) | 0 (0)
Blepharitis (Eye disorders) | 1 (1) | 0 (0)
Dry eye (Eye disorders) | 0 (0) | 1 (1)
Vision blurred (Eye disorders) | 0 (0) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 2 (2) | 4 (4)
Abdominal distension (Gastrointestinal disorders) | 2 (2) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 2 (2) | 1 (1)
Anal fissure (Gastrointestinal disorders) | 1 (1) | 0 (0)
Cheilitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colitis ischaemic (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 19 (20) | 3 (3)
Dental caries (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 6 (7) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Faeces hard (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 3 (3) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1)
Glossitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 18 (21) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 3 (3) | 1 (1)
Vomiting (Gastrointestinal disorders) | 3 (4) | 0 (0)
Asthenia (General disorders) | 1 (1) | 0 (0)
Feeling abnormal (General disorders) | 0 (0) | 1 (1)
Malaise (General disorders) | 12 (12) | 2 (2)
Peripheral swelling (General disorders) | 1 (1) | 0 (0)
Thirst (General disorders) | 19 (19) | 3 (3)
Hepatic function abnormal (Hepatobiliary disorders) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 3 (3)
Conjunctivitis (Infections and infestations) | 1 (1) | 1 (1)
Cystitis (Infections and infestations) | 0 (0) | 2 (3)
Gastroenteritis (Infections and infestations) | 2 (2) | 2 (2)
Gastroenteritis rotavirus (Infections and infestations) | 0 (0) | 1 (1)
Gingival abscess (Infections and infestations) | 1 (1) | 0 (0)
Gingivitis (Infections and infestations) | 1 (1) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 1 (1)
Hordeolum (Infections and infestations) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 2 (2)
Nasopharyngitis (Infections and infestations) | 27 (27) | 28 (30)
Oral herpes (Infections and infestations) | 1 (1) | 0 (0)
Paronychia (Infections and infestations) | 1 (1) | 0 (0)
Periodontitis (Infections and infestations) | 1 (1) | 1 (1)
Pharyngitis (Infections and infestations) | 1 (1) | 1 (1)
Tonsillitis (Infections and infestations) | 1 (1) | 0 (0)
Chillblains (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Comminuted fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 9 (10) | 7 (7)
Excoriation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Frostbite (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Ligament sprain (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Limb crushing injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Muscle injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Muscle rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Patella fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 8 (8) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 7 (7) | 1 (1)
Blood creatine phosphokinase increased (Investigations) | 1 (1) | 1 (1)
Blood creatinine increased (Investigations) | 0 (0) | 1 (1)
Blood potassium decreased (Investigations) | 1 (1) | 0 (0)
Blood potassium increased (Investigations) | 0 (0) | 2 (2)
Blood uric acid increased (Investigations) | 0 (0) | 1 (1)
Blood urine present (Investigations) | 3 (3) | 1 (1)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 3 (3)
Liver function test abnormal (Investigations) | 1 (1) | 0 (0)
White blood cell count increased (Investigations) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 9 (9) | 1 (1)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (4)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 8 (10)
Costochondritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Limb discomfort (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Myalgia intercostal (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Nodal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Periarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3)
Synovitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Tenosynovitis stenosans (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Carpal tunnel syndrome (Nervous system disorders) | 0 (0) | 1 (1)
Cerebral infarction (Nervous system disorders) | 0 (0) | 1 (1)
Cervicobrachial syndrome (Nervous system disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 2 (3) | 2 (2)
Dizziness postural (Nervous system disorders) | 1 (1) | 0 (0)
Dysgeusia (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 5 (11)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 1 (1)
Loss of consciousness (Nervous system disorders) | 1 (1) | 0 (0)
Migraine (Nervous system disorders) | 1 (1) | 0 (0)
Sciatica (Nervous system disorders) | 1 (1) | 3 (3)
Somnolence (Nervous system disorders) | 24 (24) | 6 (6)
Abulia (Psychiatric disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 3 (3) | 0 (0)
Dysuria (Renal and urinary disorders) | 2 (2) | 0 (0)
Hypertonic bladder (Renal and urinary disorders) | 1 (1) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Stress urinary incontinence (Renal and urinary disorders) | 1 (1) | 0 (0)
Urethral haemorrhage (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 1 (1) | 0 (0)
Urine flow decreased (Renal and urinary disorders) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 3 (5) | 1 (2)
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Eczema asteatotic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Haemorrhage subcutaneous (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Ingrowing nail (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Prurigo (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hot flush (Vascular disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 1 (1)
Peripheral arterial occlusive disease (Vascular disorders) | 0 (0) | 1 (1)
Varicose vein (Vascular disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days